CLINICAL TRIAL: NCT06454383
Title: A Phase 1b Study of Gemcitabine and Leflunomide in Patients With Unresectable Pancreatic Cancer
Brief Title: Gemcitabine and Leflunomide in Patients With Advanced Unresectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23540; NCI-2024-04359 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23540 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Advanced Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Specimen Handling; Cholestyramine Resin; X-Rays; Gemcitabine; Leflunomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (gemcitabine, leflunomide) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 of each cycle and leflunomide PO QD on days -3 to -1 prior to cycle 1 and days 1-28 of each cycle thereafter. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive cholestyramine PO TID for 11 days at the end of treatment in the absence of unacceptable toxicity. Patients also undergo CT, MRI, or other imaging scans as clinically indicated throughout the study, as well as blood sample collection on study and during follow up.
  Interventions: Procedure: Biospecimen Collection; Drug: Cholestyramine; Procedure: Computed Tomography; Procedure: Diagnostic Imaging; Drug: Gemcitabine; Drug: Leflunomide; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cholestyramine — Given PO
  Other Names: Cholybar; Colestyramine; Duolite AP143 Resin; Questran; Questran Light
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Diagnostic Imaging — Undergo imaging scans
  Other Names: Medical Imaging
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Leflunomide — Given PO
  Other Names: Arava; SU101
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of leflunomide in combination with gemcitabine in treating patients with pancreatic cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and cannot be removed by surgery (unresectable). Improving the effectiveness of gemcitabine without increasing side effects could lead to a greater impact for pancreatic cancer patients' survival and quality of life. Gemcitabine is commonly used as a first-line chemotherapy treatment for pancreatic cancer. Leflunomide is a drug approved for use against rheumatoid arthritis that is being looked at as a cancer treatment option. It has shown promising results when combined with gemcitabine. Giving gemcitabine in combination with leflunomide may be safe and effective in treating patients with advanced unresectable pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of gemcitabine in combination with leflunomide and determine the recommended Phase 2 dose (RP2D) of the combination.

SECONDARY OBJECTIVES:

I. To evaluate the progression-free (PFS) and overall survival (OS). II. To evaluate the overall response rate (ORR), including confirmed and unconfirmed, complete and partial response and stable disease.

III. To describe quality of life utilizing the Functional Assessment of Cancer Therapy: General (FACT-G) questionnaire.

EXPLORATORY OBJECTIVES:

I. To describe the pharmacokinetic profile of leflunomide when given in combination with gemcitabine.

II. To examine the relationship between pharmacokinetics and disease progression.

OUTLINE:

Patients receive gemcitabine intravenously (IV) over 30 minutes on days 1, 8, and 15 of each cycle and leflunomide orally (PO) once daily (QD) on days -3 to -1 prior to cycle 1 and days 1-28 of each cycle thereafter. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive cholestyramine PO three times a day (TID) for 11 days at the end of treatment in the absence of unacceptable toxicity. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), or other imaging scans as clinically indicated throughout the study, as well as blood sample collection on study and during follow up.

After completion of study treatment, patients are followed up at 30 days then up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Adult patients lacking capacity to consent may participate if they have a caretaker that could ensure oral medication compliance.
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies.

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval.
* Age: ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) ≤ 1.
* Subjects must have histologically or cytologically confirmed diagnosis of advanced unresectable pancreatic ductal adenocarcinoma (PDA).
* Measurable or evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1
* Potential patients must have plans of receiving single agent gemcitabine.
* Fully recovered from the acute toxic effects (except alopecia or neuropathy) to ≤ grade 1 to prior anti-cancer therapy.
* Without bone marrow involvement: Absolute neutrophil count (ANC) ≥ 1,500/mm^3 NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement.
* Without bone marrow involvement: Platelets ≥ 100,000/mm^3 NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement.
* Hemoglobin ≥ 9g/dL NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment unless cytopenia is secondary to disease involvement.
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 x ULN (unless has Gilbert's disease total bilirubin ≤ 3 x ULN)
* Aspartate aminotransferase (AST) ≤ 1.5 x ULN OR if liver metastases ≤ 3 x ULN
* Alanine aminotransferase (ALT) ≤ 1.5 x ULN OR if liver metastases ≤ 2 x ULN
* Creatinine ≤ 1.5 x ULN OR creatinine clearance (Cockcroft Gault) of ≥ 50 mL/min for participants with a creatinine level of > 1.5 x ULN.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of gemcitabine therapy for women and at least 3 months after the last dose of gemcitabine therapy for men, and/or undergo drug elimination of leflunomide at end of treatment until leflunomide is undetectable in the plasma.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy.
* Drugs metabolized by CYP2C8, CYP1A2, BCRP, OATP1B1/B3, and OAT3 transporters within 21 days prior to day 1 of protocol therapy.
* Herbal medications (excluding cannabidiol [CBD]).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Issues with tolerating oral medication (e.g. inability to swallow pills, malabsorption issues, ongoing nausea or vomiting).
* Positive for tuberculosis or latent tuberculosis (TB).
* Active diarrhea.
* Clinically significant uncontrolled illness.
* Active infection requiring antibiotics.
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection. (*If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable.)
* Diagnosis of Gilbert's disease.
* Prior malignancy other than carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated 5 or more years prior to study entry with no subsequent evidence of recurrence. Patients with a history of low grade (Gleason score ≤ 6 = Gleason group 1) localized prostate cancer will be eligible even if diagnosed less than 5 years prior to study entry. Other malignancies with low probability of recurrence may be allowed with PI approval.
* Females only: Pregnant or breastfeeding.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | Up to 28 days (cycle 1)
  Toxicities will be graded according to Common Terminology Criteria for Adverse Events version 5.0.
Incidence of adverse events | Up to 30 days after completion of study treatment
  Toxicities will be graded according to Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From start of protocol treatment until progression or death, and if neither event occur, the patient is at the time of last contact, assessed up to 1 year after completion of study treatment
  PFS will be estimated using the Kaplan-Meier product-limit method.
Overall survival (OS) | From start of protocol treatment until death, and if the patient is alive, the patient is censored at time of last contact, assessed up to 1 year after completion of study treatment
  OS will be estimated using the Kaplan-Meier product limit method.
Overall response rate (ORR) | Up to 1 year after completion of study treatment
  ORR will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.
Change in quality of life (QOL) | Baseline to 1 year after completion of study treatment
  Change in QOL will be measured by the Functional Assessment of Cancer Therapy: General (FACT-G) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States